CLINICAL TRIAL: NCT03618459
Title: Persistent Post-discharge Pain After Breast Surgery With Paravertebral Block: Incidence, Characteristics and Consequences
Brief Title: Post-discharge Pain After Breast-surgery Treated by Paravertebral Block
Status: Completed | Type: Observational
Sponsor: Samuele Ceruti (Other)
Collaborators: Ente Ospedaliero Cantonale, Bellinzona (Other)
Responsible Party: Sponsor-Investigator, Samuele Ceruti, Principal Investigator, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Other Study IDs: CERU-1802
Record Dates: First submitted 2018-07-26; First posted 2018-08-07 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Mastectomy, Segmental; Regional Anesthesia
Keywords: Breast surgery; Paravertebral block; Pain Control
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast-surgery patients: A consecutive cohort of adult patients undergoing breast surgery with a combined anesthesia technique, employing a thoracic single-shot paravertebral block performed before surgery. Operations performed were in all cases unilateral tumor resections, lumpectomies and mastectomies without axillary lymphadenectomy.
  Interventions: Other: Phone questionnaire

INTERVENTIONS:
Other: Phone questionnaire — Patients were contacted by phone 6 months after surgery and, after oral consent, a standardized questionnaire was administered in order to inquiry about the length and nature of post-operative pain, the incidence of post-discharge pain, its characteristics, its impact on daily life, its treatment and its rate of chronicity

SUMMARY:
Breast surgery is known being associated to a high risk of persistent post-operative pain, which has been related, among other factors, to a poorly treated acute pain. Paravertebral block has been successfully employed for anesthesia and analgesia after breast surgery, however its impact on persistent post-operative pain has rarely been investigated. Aim of this study is to assess prevalence, characteristics and consequences of post-discharge pain and its correlation to the incidence of persistent post-operative pain development in a continuous cohort of patients undergoing breast surgery with a paravertebral block.

Investigators designed a prospective, observational study on a continuous cohort of adult patients undergoing breast surgery with a standardized thoracic paravertebral block performed before general anesthesia induction. Patients were subsequently interviewed 6 months after hospital discharge in order to assess the incidence, features and duration of post-discharge pain.

DETAILED DESCRIPTION:
Breast cancer is the most frequent cancer in women, with an incidence of more than one million new cases per year. In the majority of cases surgery is part of the treatment and prognosis has progressively improved during last years. Attention is thus being increasingly focusing on these patients' quality of life and chronic postsurgical pain, defined as pain in the area of surgery lasting beyond 3 month from the operation, has emerged as a frequent long-term complication, with prevalence up to 60%. This often-disabling condition has been shown to significantly affect cancer survivors' quality of life and to have a heavy economic impact on the healthcare system.

Many potential risk factors have been proposed for the development of chronic post-breast surgery pain. A Cochrane systematic review has addressed the role of regional anesthesia in preventing the development of chronic postoperative pain, suggesting that "paravertebral block may reduce the pain after breast cancer surgery in about one out every five women treated", these results being however weakened by the often poor quality and inadequate power of the studies available. Many predictors of chronic postoperative pain have been identified, one of them being a poorly treated acute pain; in this perspective, regional anesthesia could possibly play a role in preventing nervous system remodeling with resultant hyperalgesia, allodynia and sustained wound pain.

Even if chronic postoperative pain has been progressively recognized as an issue after breast cancer surgery, its link to poorly treated acute postoperative pain and post-discharge pain (PDP) has been poorly investigated. Single shot paravertebral block is an effective technique to provide both anesthesia and good analgesia after breast surgery, but its benefits duration is still debated.

ELIGIBILITY:
Inclusion Criteria:

* female sex
* 18 years or greater
* elective breast surgery (tumor resection, mastectomy, lumpectomy)
* local regional anesthesia

Exclusion Criteria:

* patients refusal,
* general contraindications to regional anesthesia,
* the inability to perform a complete block
* diagnosed COPD or other respiratory diseases,
* ASA score risk greater than 3.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A consecutive cohort of adult patients undergoing breast surgery with a combined anesthesia technique, employing a thoracic single-shot paravertebral block performed before surgery. Operations performed were in all cases unilateral tumor resections, lumpectomies and mastectomies without axillary lymphadenectomy.
Sampling Method: Non-Probability Sample
Enrollment: 244 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Post-discharge pain | 6 months post-surgery
  Primary endpoint of this study is to assess the incidence of post-discharge pain in a cohort of patients undergoing breast surgery with a single shot thoracic paravertebral block.

SECONDARY OUTCOMES:
Pain characteristics | 6 months post-surgery
  Secondary endpoints is to characterize this post-discharge pain in terms of pain characteristics, evaluated by Numerical Rating Scale (NRS, from 0 intended as no pain, to 10 as maximal pain), on patient daily life after discharge home.
Pain impact | 6 months post-surgery
  Secondary endpoints is to characterize this post-discharge pain in terms of pain impact on patient daily life after discharge home, intended as capable to impact especially on a) work, b) leisure or c) sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Luciano Anselmi, MD, Study Chair — Ente Ospedaliero Cantonale, Bellinzona; Andrea Saporito, MD, Principal Investigator — Ente Ospedaliero Cantonale, Bellinzona; José Aguirre, MD, Study Director — Balgrist
Locations (1):
- Andrea Saporito MD, Bellinzona, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cronin-Fenton DP, Norgaard M, Jacobsen J, Garne JP, Ewertz M, Lash TL, Sorensen HT. Comorbidity and survival of Danish breast cancer patients from 1995 to 2005. Br J Cancer. 2007 May 7;96(9):1462-8. doi: 10.1038/sj.bjc.6603717. Epub 2007 Apr 3. PMID 17406360
- [Result] Andersen KG, Kehlet H. Persistent pain after breast cancer treatment: a critical review of risk factors and strategies for prevention. J Pain. 2011 Jul;12(7):725-46. doi: 10.1016/j.jpain.2010.12.005. Epub 2011 Mar 24. PMID 21435953
- [Result] Macdonald L, Bruce J, Scott NW, Smith WC, Chambers WA. Long-term follow-up of breast cancer survivors with post-mastectomy pain syndrome. Br J Cancer. 2005 Jan 31;92(2):225-30. doi: 10.1038/sj.bjc.6602304. PMID 15655557
- [Result] Peuckmann V, Ekholm O, Rasmussen NK, Groenvold M, Christiansen P, Moller S, Eriksen J, Sjogren P. Chronic pain and other sequelae in long-term breast cancer survivors: nationwide survey in Denmark. Eur J Pain. 2009 May;13(5):478-85. doi: 10.1016/j.ejpain.2008.05.015. Epub 2008 Jul 16. PMID 18635381
- [Result] Blyth FM, March LM, Brnabic AJ, Cousins MJ. Chronic pain and frequent use of health care. Pain. 2004 Sep;111(1-2):51-8. doi: 10.1016/j.pain.2004.05.020. PMID 15327808
- [Result] Blyth FM, March LM, Cousins MJ. Chronic pain-related disability and use of analgesia and health services in a Sydney community. Med J Aust. 2003 Jul 21;179(2):84-7. doi: 10.5694/j.1326-5377.2003.tb05441.x. PMID 12864718
- [Result] Andreae MH, Andreae DA. Local anaesthetics and regional anaesthesia for preventing chronic pain after surgery. Cochrane Database Syst Rev. 2012 Oct 17;10:CD007105. doi: 10.1002/14651858.CD007105.pub2. PMID 23076930
- [Result] Schreiber KL, Martel MO, Shnol H, Shaffer JR, Greco C, Viray N, Taylor LN, McLaughlin M, Brufsky A, Ahrendt G, Bovbjerg D, Edwards RR, Belfer I. Persistent pain in postmastectomy patients: comparison of psychophysical, medical, surgical, and psychosocial characteristics between patients with and without pain. Pain. 2013 May;154(5):660-668. doi: 10.1016/j.pain.2012.11.015. Epub 2012 Dec 5. PMID 23290256
- [Result] Staud R. Peripheral pain mechanisms in chronic widespread pain. Best Pract Res Clin Rheumatol. 2011 Apr;25(2):155-64. doi: 10.1016/j.berh.2010.01.010. PMID 22094192
- [Result] Mejdahl MK, Andersen KG, Gartner R, Kroman N, Kehlet H. Persistent pain and sensory disturbances after treatment for breast cancer: six year nationwide follow-up study. BMJ. 2013 Apr 11;346:f1865. doi: 10.1136/bmj.f1865. PMID 23580693
- [Derived] Saporito A, Aguirre J, Borgeat A, Perren A, Anselmi L, Poggi R, Minotti B, Cafarotti S, La Regina D, Ceruti S. Persistent postdischarge pain and chronic postoperative pain after breast cancer surgery under general anesthesia and single-shot paravertebral block: incidence, characteristics and impact on quality of life and healthcare costs. J Pain Res. 2019 Apr 16;12:1193-1199. doi: 10.2147/JPR.S195702. eCollection 2019. PMID 31114301